CLINICAL TRIAL: NCT03511599
Title: A Randomized, Placebo-controlled, Crossover Trial of D-cycloserine Repetitive Transcranial Magnetic Stimulation Plasticity Enhancement in the Motor System of Individuals With Major Depressive Disorder.
Brief Title: Cycloserine rTMS Plasticity Augmentation in Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: REB18-0604
Record Dates: First submitted 2018-04-18; First posted 2018-04-30 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Cycloserine; Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- D-Cycloserine (Experimental): Participants will ingest a capsule containing 100mg of the antibiotic d-cycloserine. Their baseline motor evoked potentials (MEP) will be recorded for 30 minutes prior to receiving theta-burst stimulation (TBS; a patterned stimulation) to the motor cortex and change in MEP amplitude will be measured following stimulation up to 90 minutes later and then once again the following morning (16 hours later).
  Interventions: Drug: Cycloserine; Device: Transcranial Magnetic Stimulation
- Placebo (Active Comparator): Participants will ingest a capsule identical to the study medication, however this capsule will contain a placebo.Their baseline motor evoked potentials (MEP) will be recorded for 30 minutes prior to receiving theta-burst stimulation (TBS; a patterned stimulation) to the motor cortex and change in MEP amplitude will be measured following stimulation up to 90 minutes later and then once again the following morning (16 hours later).
  Interventions: Device: Transcranial Magnetic Stimulation; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Cycloserine — Cycloserine 100mg
  Arms: D-Cycloserine
Device: Transcranial Magnetic Stimulation — Single-pulse transcranial magnetic stimulation and theta-burst stimulation
Drug: Placebo Oral Tablet — Placebo tablet matched to cycloserine tab
  Arms: Placebo

SUMMARY:
Transcranial magnetic stimulation (rTMS) is an investigational and therapeutic modality that impacts the connection strength between neurons by delivering patterned energy. In response to this patterned energy neurons fire and adapt by changing their connection strengths. This change in connection strengths is believed to be the underlying mechanism whereby this intervention has therapeutic benefit for this intervention in conditions such as depression. The purpose of this study is to test a means of enhancing the effect of rTMS using a medication (cycloserine) that has been shown to augment and stabilize activity dependent neuronal changes. The investigators wish to use the motor system, where the associated muscle response to brain stimulation can be measured, to probe activity dependent changes in connection strength between neurons.

DETAILED DESCRIPTION:
This randomized, placebo-controlled, crossover trial will enroll 12 participants with Major Depressive Disorder. In one arm of the study, participants will randomly receive either 100mg of d-cycloserine (DCS, an antibiotic) or a placebo capsule, and participants will receive the other intervention one week later.

1. We will recruit 12 participants aged 18-60 through community advertisement, carefully screened for exclusion factors related to rTMS and DCS.
2. After screening, participants will come to the lab for a semi-structured interview involving the MINI-International Neuropsychiatric Interview for confirmation of the diagnosis of depression, and the absence of substance use disorders, absence of psychosis, and absence of bipolar disorder. The severity of their depressive symptoms will be quantified with the semi-structured clinical instrument Hamilton Depression Rating Scale, and participants will be retained in the study if their score is ≥15, indicating moderate severity. Finally, the antidepressant treatment history will be collected using the Antidepressant Treatment History Form.
3. Eligible participants will be randomly assigned by random number sequence with allocation concealment to one of two first arms of the crossover study: a) placebo-DCS 100mg and b) DCS 100mg-placebo.
4. Participants will complete the QIDS-SR (Quick Inventory of Depressive Symptoms-Self Report), the MDQ (Mood Disorders Questionnaire), the BAI (Beck Anxiety Inventory), and the STAI (State Trait Anxiety Inventory). Participants will report their perception of physical symptoms (potential side effects) in the 7 days before participating in the study taking the randomized capsule (Toronto Side Effects Scale - 1 Week).
5. Participants will take their blinded capsule at least 30 minutes prior to TBS (we anticipate that it will take approximately 30 minutes to do steps 5-7).
6. Electromyographic (EMG) electrodes will be positioned over the first dorsal interosseous (FDI) bilaterally. These are non-invasive electrodes that use an adhesive to stick to the skin.
7. Using neuronavigation in conjunction with an atlas brain, the M1 hand strip will be localized using single pulse TMS (MagPro X100).
8. Motor evoked potentials are measurements of muscle activation, in this case in response to TMS stimulation of the brain. We will use single pulse TMS to record the magnitude of responses. As a baseline, we will collect twenty single-pulse (120% resting motor threshold (RMT), 0.25Hz) MEPs every 5 minutes for the 15 minutes preceding TBS rTMS.
9. We will characterize a stimulus response curve by delivering single pulse TMS at stimulation intensities ranging from 100-150% of resting motor threshold in random order.
10. TBS rTMS will be applied to the FDI 'hotspot'. TBS consists of 2s trains every 10s. Trains are composed of 3 pulses at 50Hz, 200ms intervals, 80% RMT. Total time 190s and 600 pulses.
11. After TBS, twenty MEPs will be acquired (single pulse, 120% RMT, 0.25Hz) every 5 minutes for the first 30 minutes, at 60 minutes, at 90 minutes, and at 16Hrs (the following morning).
12. At the 90 minute and 16 Hrs timepoints, we will characterize stimulus response curves (MEPs at stimulus intensities ranging from 100-150% resting motor threshold presented in random order).
13. Participants will report their perception of side effects since taking the randomized capsule (Toronto Side Effects Scale - 1 Day). Participants will be asked if they believe they received the study medication or placebo in this first phase of the crossover trial.

This study involves a crossover design, therefore after a minimum of 7 days, participants will return to the laboratory to repeat steps 4-13 with the other arm of the trial (i.e. participants who initially received the active study medication will instead receive the placebo, and the converse).

ELIGIBILITY:
Inclusion Criteria:

1. Individuals currently experiencing a major depressive episode. 1.1 As determined by the MINI-International Neuropsychiatric Interview 1.2 Moderate severity, as indicated by a Hamilton Depression Rating Scale score of ≥15.

   1.3 Be willing to remain on a stable medication regimen for 4 weeks prior the study and during the study
2. Aged 18-60

Exclusion Criteria:

1. Pregnancy
2. Lactation
3. Epilepsy
4. Previous Stroke
5. Current Renal Disease
6. Current Liver Disease
7. Current Alcohol Use Disorder
8. Inability to refrain from alcohol use for 24 hours prior to each session and following each session.
9. Allergy to antibiotics
10. Use of isoniazid, ethionamide, or bupropion
11. History of psychosis
12. History of bipolar disorder
13. Family history of bipolar disorder
14. Intracranial metallic objects (dental hardware is not an exclusionary criteria)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2021-04-21 (Actual)

PRIMARY OUTCOMES:
Motor evoked potential amplitude | Baseline versus 90 minutes following theta-burst stimulation.
  Change in the (electrical) amplitude of muscle responses to stimulation of the motor cortex will be recorded from the first dorsal interosseous muscle of the hand.

SECONDARY OUTCOMES:
Motor evoked potential dose-response curve | Baseline versus 90 minutes after theta-burst stimulation.
  Motor evoked potentials at stimulus intensities ranging from 100-150% resting motor threshold, presented at random order.
Motor evoked potential dose-response curve | Baseline versus 16 hours following theta-burst stimulation.
  Motor evoked potentials at stimulus intensities ranging from 100-150% resting motor threshold, presented at random order.
Motor evoked potential amplitude | Baseline and the evolution over 90 minutes following theta-burst stimulation.
  Change in the (electrical) amplitude of muscle responses to stimulation of the motor cortex will be recorded from the first dorsal interosseous muscle of the hand.

OTHER OUTCOMES:
Safety outcomes | Through study completion, on average 2 weeks.
  Adverse events will be tracked and recorded
Side effects | Baseline and 16 hours post-stimulus for both arms of the crossover study.
  Side effects will be tracked with the Toronto Side Effects Questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
There will be no sharing of IPD.